CLINICAL TRIAL: NCT00227253
Title: The Chromosome 18 Clinical Research Center
Brief Title: Chromosome 18 Clinical Research Center
Acronym: Chromosome18
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Other Study IDs: Chromosome 18; 5M01RR001346 (NIH)
Record Dates: First submitted 2005-09-14; First posted 2005-09-27 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Chromosome Aberrations; Growth Hormone Deficiency; Hypomyelination
Keywords: Phenotype; Growth; Genotype; Chromosome 18
MeSH Terms: conditions — Chromosome Aberrations; Dwarfism, Pituitary | interventions — Thyroid (USP)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood specimens are collected from study participant and both biological parents if available and are processed for DNA and to establish cell lines
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Determination of growth hormone status — Growth hormone stimulating testing using Arginine and Clonidine, Corticotrophin releasing hormone stimulation test
Procedure: Measurement of growth, thyroid and sex hormone levels — Gonadotrophin releasing hormone stimulation test Thyroid testing - T4, TSH, T3 uptake, and anti-thyroidal antibodies baseline sample - no medication administered
Procedure: Behavior and neuropsychometric evaluations — evaluation by neuropsychologist, standardized testing geared to study participant's age, abilities and past medical history
Procedure: Audiological and ear, nose and throat examination — neurotological exam, behavioral audiometry, immittance audiometry, assessment of the function of the inner ear using otoacoustic emissions, Auditory brain responses
Procedure: Magnetic resonance imaging of the brain — MRI of the brain - standard clinical procedure
Procedure: Dysmorphology evaluation — Genetic evaluation with picture and measurements, physical exam
Procedure: Neurology examination — physical examination including observation of balance, coordination and reflexes.
Procedure: Dental evaluation — Visual detal inspection with panorex X-ray of the entire mouth
Procedure: Speech pathology evaluation — Standardized speech & language tests and naturalistic assessment procedures.
Procedure: Psychiatric evaluation — Psychiatric interview about history of psychiatric and medical illnesses, family psychiatric and medical history, demographic info also obtained
Procedure: Orthopedic evaluation — Physical exam by orthopedic surgeon and a dysplasia series of radiographs including AP and lateral radiographics of the feet, APs of the knees, pelvis, thoracic lumbar spine and chest, laterals of thoracic lumbar and cervical spine, lateral of the skull, AP and lateral of the forearm, bone age evaluation with radiograph of left hand
Procedure: Ophthalmologic evaluation — exam will determine visual acuity using one of the following: Snellen chart, Allen acuity, target acuity, optokinetic nystagmus (OKN), or Teller acuity depending on study participants ability level. Motility/alignment will also be determined using cover/uncover test. Pupils examined using slit lamp. Dilated fundus exam and cycloplegic refraction which will require dilating drops in both eyes. Cyclogen 1% and NeuSynephrine 2.5% are using. In children less than 6 months old, less potent mydriatrics and cycloplegics are used Cyclogel 0.5% or Tropicamide 1%. Intraocular pressure will be measured in adults and cooperative teens using applanation tonometry. A topical anesthetic will be used to perform this measurement.
Procedure: Gastrointestinal evaluation — physical exam and medical history by board certified gastroenterologist.

SUMMARY:
Our vision, that of the researchers at the University of Texas Health Science Center at San Antonio, is that every person with a chromosome 18 abnormality will have an autonomous and healthy life. Our mission is to provide families affected by chromosome 18 abnormalities with comprehensive medical and educational information. Our goals are to provide definitive medical and education resources for the families of individuals with chromosome 18 abnormalities; perform and facilitate groundbreaking clinical and basic research relating to the syndromes of chromosome 18; and to provide treatments to help these individuals overcome the effects of their chromosome abnormality.

DETAILED DESCRIPTION:
Protocol Summary:

The hypotheses are:

1. growth hormone (GH) deficiency in children with chromosome 18 deletions is accompanied by cognitive and microstructural abnormalities of the brain that can be ameliorated by GH treatment; and
2. the physical and behavioral findings in individuals with abnormalities of chromosome 18 are due to the genes that present in a non-diploid number.

Therefore, correlation of the physical and behavioral findings with the extent of the deletion will help identify the genes involved. An understanding of the molecular mechanisms of the phenotype will provide the insight necessary to devise appropriate therapies.

Our goals are:

1. to be the international medical and education resource for the families of individuals with chromosome 18 abnormalities;
2. to perform and facilitate both clinical and basic research relating to the disorders of chromosome 18; and
3. to devise treatments to help these individuals overcome the negative effects of their chromosome abnormality.

To attain these goals, the study has the following specific aims:

1. perform genotypic molecular analysis on the DNA of the subjects and their biological parents to determine the genotype of the affected individual;
2. gather comprehensive clinical data on individuals with chromosome 18 abnormalities including:

   1. determination of growth hormone levels;
   2. measurement of corticotrophin, thyroid and sex hormones;
   3. psychiatric and neuropsychological evaluations;
   4. audiology and ENT testing;
   5. brain MRI scan;
   6. genetic dysmorphology examination;
   7. neurology exam;
   8. dental exam;
   9. speech pathology evaluation;
   10. gastrointestinal exam;
   11. orthopedic exam;
   12. ophthalmology exam.

The phenotypical assessment will be longitudinal; therefore, the participants will have a wide age range. This extensive range plus the fact that some participants will be assessed multiple times means that not all components of the clinical studies will be appropriate for every subject at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of Chromosome 18 or be the parent/guardian of a child with Chromosome 18
* Subject must be at least one year of age to participate in the clinical examination aspect of the study (due to issues of venous access and blood volume required to complete studies)
* General health status: good

Exclusion Criteria:

* Pregnant women
* Dead fetuses
* Prisoners
* Non-viable neonates or neonates of uncertain viability

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Must have a confirmed diagnosis of Chromosome 18 or be the parent/guardian of a child with Chromosome 18
  * Subject must be at least one year of age to participate in the clinical examination aspect of the study (due to issues of venous access and blood volume required to complete studies)
  * General health status: good
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 1993-09; Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Primary | Ongoing
  Provide definitive medical and education resources for the families of individuals with chromosome 18 abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Jannine D. Cody, Ph.D., Principal Investigator — The University of Texas Health Science Center at San Antonio; Jonathan Gelfond, M.D., Ph.D., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - University Health Systems Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Result] Cody JD, Semrud-Clikeman M, Hardies LJ, Lancaster J, Ghidoni PD, Schaub RL, Thompson NM, Wells L, Cornell JE, Love TM, Fox PT, Leach RJ, Kaye CI, Hale DE. Growth hormone benefits children with 18q deletions. Am J Med Genet A. 2005 Aug 15;137(1):9-15. doi: 10.1002/ajmg.a.30848. PMID 16007630
- [Result] Lancaster JL, Cody JD, Andrews T, Hardies LJ, Hale DE, Fox PT. Myelination in children with partial deletions of chromosome 18q. AJNR Am J Neuroradiol. 2005 Mar;26(3):447-54. PMID 15760848
- [Result] Kochunov P, Lancaster J, Hardies J, Thompson PM, Woods RP, Cody JD, Hale DE, Laird A, Fox PT. Mapping structural differences of the corpus callosum in individuals with 18q deletions using targetless regional spatial normalization. Hum Brain Mapp. 2005 Apr;24(4):325-31. doi: 10.1002/hbm.20090. PMID 15704090
- [Result] Schaub RL, Hale DE, Rose SR, Leach RJ, Cody JD. The spectrum of thyroid abnormalities in individuals with 18q deletions. J Clin Endocrinol Metab. 2005 Apr;90(4):2259-63. doi: 10.1210/jc.2004-1630. Epub 2005 Jan 25. PMID 15671099
- [Result] Cody JD, Hale DE. Precision in phenotyping and genotyping. Am J Med Genet A. 2004 Dec 15;131(3):313. doi: 10.1002/ajmg.a.30263. No abstract available. PMID 15540176
- [Result] Gunn SR, Mohammed M, Reveles XT, Viskochil DH, Palumbos JC, Johnson-Pais TL, Hale DE, Lancaster JL, Hardies LJ, Boespflug-Tanguy O, Cody JD, Leach RJ. Molecular characterization of a patient with central nervous system dysmyelination and cryptic unbalanced translocation between chromosomes 4q and 18q. Am J Med Genet A. 2003 Jul 1;120A(1):127-35. doi: 10.1002/ajmg.a.20026. PMID 12794705
- [Result] Schaub RL, Reveles XT, Baillargeon J, Leach RJ, Cody JD. Molecular characterization of 18p deletions: evidence for a breakpoint cluster. Genet Med. 2002 Jan-Feb;4(1):15-9. doi: 10.1097/00125817-200201000-00003. PMID 11839953
- [Result] Schaub RL, Cody JD, Hale DE. Growth disorders in the chromosome 18 syndromes. Highlights 9:3-5, 2001
- [Result] Hermesch CB, Cody JT, Cody JD. Dental caries history in nine children with chromosome 18p deletion syndrome. Spec Care Dentist. 2000 Mar-Apr;20(2):53-5. doi: 10.1111/j.1754-4505.2000.tb01143.x. PMID 11203878
- [Result] Hale DE, Cody JD, Baillargeon J, Schaub R, Danney MM, Leach RJ. The spectrum of growth abnormalities in children with 18q deletions. J Clin Endocrinol Metab. 2000 Dec;85(12):4450-4. doi: 10.1210/jcem.85.12.7016. PMID 11134092
- [Result] Cody JD, Reveles XT, Hale DE, Lehman D, Coon H, Leach RJ. Haplosufficiency of the melancortin-4 receptor gene in individuals with deletions of 18q. Hum Genet. 1999 Nov;105(5):424-7. doi: 10.1007/s004390051125. PMID 10598807
- [Result] Wang Z, Cody JD, Leach RJ, O'Connell P. Gene expression patterns in cell lines from patients with 18q- syndrome. Hum Genet. 1999 Jun;104(6):467-75. doi: 10.1007/s004390050989. PMID 10453734
- [Result] Cody JD, Ghidoni PD, DuPont BR, Hale DE, Hilsenbeck SG, Stratton RF, Hoffman DS, Muller S, Schaub RL, Leach RJ, Kaye CI. Congenital anomalies and anthropometry of 42 individuals with deletions of chromosome 18q. Am J Med Genet. 1999 Aug 27;85(5):455-62. doi: 10.1002/(sici)1096-8628(19990827)85:53.0.co;2-z. PMID 10405442
- [Result] Brkanac Z, Cody JD, Leach RJ, DuPont BR. Identification of cryptic rearrangements in patients with 18q- deletion syndrome. Am J Hum Genet. 1998 Jun;62(6):1500-6. doi: 10.1086/301854. PMID 9585582
- [Result] Keppler-Noreuil KM, Carroll AJ, Finley SC, Descartes M, Cody JD, DuPont BR, Gay CT, Leach RJ. Chromosome 18q paracentric inversion in a family with mental retardation and hearing loss. Am J Med Genet. 1998 Apr 13;76(5):372-8. doi: 10.1002/(sici)1096-8628(19980413)76:53.0.co;2-p. PMID 9556294
- [Result] Cody JD, Hale DE, Brkanac Z, Kaye CI, Leach RJ. Growth hormone insufficiency associated with haploinsufficiency at 18q23. Am J Med Genet. 1997 Sep 5;71(4):420-5. PMID 9286448
- [Result] Gay CT, Hardies LJ, Rauch RA, Lancaster JL, Plaetke R, DuPont BR, Cody JD, Cornell JE, Herndon RC, Ghidoni PD, Schiff JM, Kaye CI, Leach RJ, Fox PT. Magnetic resonance imaging demonstrates incomplete myelination in 18q- syndrome: evidence for myelin basic protein haploinsufficiency. Am J Med Genet. 1997 Jul 25;74(4):422-31. doi: 10.1002/(sici)1096-8628(19970725)74:43.0.co;2-k. PMID 9259379
- [Result] Cody JD, Pierce JF, Brkanac Z, Plaetke R, Ghidoni PD, Kaye CI, Leach RJ. Preferential loss of the paternal alleles in the 18q- syndrome. Am J Med Genet. 1997 Mar 31;69(3):280-6. doi: 10.1002/(sici)1096-8628(19970331)69:33.0.co;2-n. PMID 9096757
- [Result] Ghidoni PD, Hale DE, Cody JD, Gay CT, Thompson NM, McClure EB, Danney MM, Leach RJ, Kaye CI. Growth hormone deficiency associated in the 18q deletion syndrome. Am J Med Genet. 1997 Mar 3;69(1):7-12. doi: 10.1002/(sici)1096-8628(19970303)69:13.0.co;2-p. PMID 9066876
- [Result] Carter E, Heard P, Hasi M, Soileau B, Sebold C, Hale DE, Cody JD. Ring 18 molecular assessment and clinical consequences. Am J Med Genet A. 2015 Jan;167A(1):54-63. doi: 10.1002/ajmg.a.36822. Epub 2014 Oct 22. PMID 25339348
- [Result] Cody JD, Sebold C, Heard P, Carter E, Soileau B, Hasi-Zogaj M, Hill A, Rupert D, Perry B, O'Donnell L, Gelfond J, Lancaster J, Fox PT, Hale DE. Consequences of chromsome18q deletions. Am J Med Genet C Semin Med Genet. 2015 Sep;169(3):265-80. doi: 10.1002/ajmg.c.31446. Epub 2015 Aug 3. PMID 26235940
- [Result] Cody JD, Hale DE. Making chromosome abnormalities treatable conditions. Am J Med Genet C Semin Med Genet. 2015 Sep;169(3):209-15. doi: 10.1002/ajmg.c.31447. PMID 26351122
- [Result] Hasi-Zogaj M, Sebold C, Heard P, Carter E, Soileau B, Hill A, Rupert D, Perry B, Atkinson S, O'Donnell L, Gelfond J, Lancaster J, Fox PT, Hale DE, Cody JD. A review of 18p deletions. Am J Med Genet C Semin Med Genet. 2015 Sep;169(3):251-64. doi: 10.1002/ajmg.c.31445. Epub 2015 Aug 6. PMID 26250845
- [Result] Sebold C, Soileau B, Heard P, Carter E, O'Donnell L, Hale DE, Cody JD. Whole arm deletions of 18p: medical and developmental effects. Am J Med Genet A. 2015 Feb;167A(2):313-23. doi: 10.1002/ajmg.a.36880. Epub 2015 Jan 14. PMID 25586871
- [Result] Cody JD, Hasi M, Soileau B, Heard P, Carter E, Sebold C, O'Donnell L, Perry B, Stratton RF, Hale DE. Establishing a reference group for distal 18q-: clinical description and molecular basis. Hum Genet. 2014 Feb;133(2):199-209. doi: 10.1007/s00439-013-1364-6. Epub 2013 Oct 5. PMID 24092497
- See also: Click here for more information about this study: The Chromosome 18 Clinical Research Center — https://wp.uthscsa.edu/chrome-18/
- See also: The Chromosome 18 Registry & Research Society is a lay advocacy organization composed primarily of the parents of individuals with one of the chromosome 18 abnormalities. — http://www.chromosome18.org